CLINICAL TRIAL: NCT06114537
Title: Randomized Clinical Trial to Evaluate the Efficacy of Acetazolamide for the Treatment of Cystoid Fluid Collections in Retinoschisis: The AXIS Trial
Brief Title: The AXIS Study: the Efficacy of Acetazolamide for the Treatment of Cystoid Fluid Collections in Retinoschisis
Acronym: AXIS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Camiel J. F. Boon, Principal Investigator and Clinical Professor, Amsterdam UMC, location AMC
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL80249.018.22
Record Dates: First submitted 2023-10-24; First posted 2023-11-02 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Retinoschisis
Keywords: X-Linked Retinoschisis; X-Linked Juvenile Retinoschisis
MeSH Terms: conditions — Retinoschisis | interventions — Acetazolamide

STUDY DESIGN:
Intervention Model Description: Patients will be randomized into the treatment group or the control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment group (Experimental): Patients in the treatment group receives twice daily a 250mg tablet acetazolamide for 16 weeks. At week 16, depending on the results, the treated group will stop the treatment or continue with a lower dose twice daily a 125mg tablet acetazolamide for 4 weeks. At week 20, depending on the results, the initial treated group will continue with twice daily a 125mg tablet or go back to twice daily a 250mg tablet acetazolamide till week 32.
  Interventions: Drug: Acetazolamide
- Control Group (No Intervention)

INTERVENTIONS:
Drug: Acetazolamide — The used intervention in this study is acetazolamide, which belongs to a class of drugs known as carbonic anhydrase inhibitors and has been used with other medications to treat high ocular pressure due to certain types of glaucoma
  Patients in the treatment group will receive 250 milligrams of oral acetazolamide twice daily for 16 weeks.
  Patients randomized to the treatment group will switch to 125 milligrams of oral acetazolamide twice daily for another four weeks when the central foveal thickness (CFT) on OCT is reduced by ≥25% at the evaluation visit at 16 weeks after the baseline visit. These patients will continue with this dose till the end of the study when the CFT on OCT is stable or further reduced. If the CFT on OCT has increased, they switch back to 250 milligrams of oral acetazolamide twice daily for another 12 weeks.
  Other Names: Diamox
  Arms: Treatment group

SUMMARY:
X-linked retinoschisis (XLRS) is a rare hereditary eye disease that causes irreversible vision loss in boys and young men. This disease occurs in 1 in 10,000-30,000. This inherited condition is caused by pathogenic variants in a single gene, namely the Retinoschisin 1 (RS1). This gene encodes the retinoschisin protein. Pathological variants of retinoschisin lead to loss of retinal integrity, resulting in the characteristic cystoid fluid collections (CFC). From a young age, XLRS patients experience a gradual deterioration of vision. In middle-aged patients however, XLRS may be associated with macular atrophy because of the confluence of the cystoid lesions. No permanent treatment is yet available for XLRS patients. Currently, two different phase I/II studies are investigating the safety and effectivity of subretinal gene therapy. To create optimal retinal condition before gene therapy, CFC, a hallmark of XLRS, should not be present. Topical and oral carbonic anhydrase II inhibitors are used to combat CFC. This drug is still off-label prescribed for various hereditary retinal dystrophies. Consequently, there is no treatment regimen for prescribing acetazolamide to XLRS patients. A thorough understanding of the safety and efficacy of acetazolamide in reducing the central foveal thickness in XLRS patients is required before applying future gene therapy.

The proposed study is a investigator-initiated, single-center, prospective, experimental study consisting of seven visits at 2, 4, 12, 16, 20 and 32 weeks after the baseline evaluation visit. During each visit, participants will perform several ophthalmological measurements. In this study, participants with XLRS will be randomized into either a treatment or control group. The null-hypothesis of this study is that acetazolamide effectively reduces the central foveal thickness in patients with XLRS and significantly improves their visual function. The alternative hypothesis is that acetazolamide reduces not effectively the central foveal thickness in patients with XLRS and has no significant impact on their visual function. Treatment success will be based not only on anatomical improvement, but also on functional endpoints, which are most important from a patient's perspective. The study will last 32 weeks per participant. Each participant will come physically for seven visits. The whole study will last for max. 24 months. The examinations and number of visits are reduced to a minimum. In contrast to clinical care, the participants receive examinations that consist of a more extensive measurement of visual acuity, microperimetry and a questionnaire. These extra examinations are required to evaluate the functional vision-related endpoints of the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with XLRS with cystoid fluid collections involving the fovea confirmed on SD- OCT
* are willing to undergo ophthalmic examinations at seven separate occasions;
* have no visual dysfunction that is also significantly associated with other ocular diseases besides XLRS (e.g., glaucoma, perforating trauma);
* have no known (non-)ocular disease/disorder which may influence the results of the measurements.

Exclusion Criteria:

* Severe hepatic impairment
* Severe renal insufficiency
* Sodium and Potassium Depletion
* Addison's disease
* Hyperchloremic Acidosis
* Cor pulmonale
* Chronic non-congestive angle-closure glaucoma
* Usage of acetazolamide
* Known allergy or intolerance for ocular anesthetic eye drops oxybuprocaine 0.4% or mydriatics tropicamide 0.5% and/or phenylephrine 5%;

Min Age: 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2023-01-20 (Actual); Primary Completion 2024-09-13 (Actual); Study Completion 2024-09-13 (Actual)

PRIMARY OUTCOMES:
Macular structure as assessed by spectral domain optical coherence tomography | Change from baseline to Week 32
  Change in Central subfield thickness on spectral domain optical coherence tomography (SD-OCT).

SECONDARY OUTCOMES:
Visual acuity as assessed by low-luminance visual acuity | Change from baseline to Week 32
  Change in low luminance visual acuity (LLVA)
Visual function as assessed by microperimetry | Change from baseline to Week 32
  Change in microperimetry.
Subject-reported visual function as assessed by the Michigan Retinal Degeneration Questionnaire (MRDQ). | Change from baseline to Week 32
  Change in the functional (dis)ability score, theta score (θ), in the measured trait or domain. Θ is centred at the mean trait level of the patient population of the developers with a variance of 1, and extreme Θ-values -3 and + 3 indicate lowest and highest visual disability respectively of each patients.
Absence of cystoid fluid collections on OCT scan | At evaluation visits during study (assessed up to 32 weeks)
  Absence of cystoid fluid collections on OCT scan
Visual acuity as assessed by best-corrected visual acuity | Change from baseline to Week 32
  Change in in best-corrected visual acuity (BCVA).

CONTACTS AND LOCATIONS:
Overall Officials: Camiel JF Boon, Prof. dr., Principal Investigator — Amsterdam UMC
Locations (1):
- Amsterdam University Medical Centers, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No